CLINICAL TRIAL: NCT03682809
Title: Evaluation of Systane Complete for the Treatment of Contact Lens Discomfort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Southern College of Optometry (Other); Lindenhurst Eye Physicians & Surgeons, PC (Other); Alcon Research (Industry)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000522017
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Contact Lens Discomfort; Dry Eye
Keywords: Artificial Tears; Systane Complete; Contact Lens Discomfort; Dry Eye; Daily Disposable Contact Lenses
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: One group will be randomized Systane Complete, and one group will be randomized to no treatment.
Who Masked: Participant, Investigator
Masking Description: The patients who are randomized to Systane Complete will be masked to the brand of the artificial tears.
  There will be a masked examiner who does not know the subject's study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systane Complete (Experimental): Subjects randomized to this group will be asked to use Systane Complete once before and after contact lens use.
  Interventions: Drug: Systane Complete
- No Treatment (No Intervention): Subjects randomized to this group will not receive a treatment.

INTERVENTIONS:
Drug: Systane Complete — Systane Complete is an artificial tear indicated for patients who have evaporative, aqueous deficient, or mixed dry eye.
  Arms: Systane Complete

SUMMARY:
Clinicians commonly use artificial tears off label for treating contact lens (CL) discomfort and the dry eye associated with CLs because new artificial tear formulations have the potential to outperform the available CL rewetting drops. While off-label, McDonald et al. have previously shown that using a common artificial tear, Systane Ultra, before and after CL use is an effective means for treating daily disposable CL wears who have CL discomfort. Recently, a new formulation of artificial tears, Systane Complete, was released to the market. Systane Complete is a unique formulation that has combined elements from both Systane Ultra (indicated for aqueous deficient dry eye) and Systane Balance (indicated for evaporative dry eye) to create an artificial tear with an indication for aqueous deficient, evaporative, and mixed (both aqueous deficient and evaporative) dry eye. Thus, the goal of this study is to determine in a randomized clinical trial if Systane Complete is able to effectively improve the symptoms of patients who have CL discomfort.

DETAILED DESCRIPTION:
Soft contact lenses (CL) are the most common CL modality with over 140 million users world. Despite many improvements in CL materials and solutions, the advent of daily disposable CLs, and the addition of rewetting drops to improve CL comfort, research has shown that between 21% to 64% of CL wearers permanently discontinue CL use because of eye discomfort. Contact Lens Discomfort (CLD) as defined by the Tear Film and Ocular Surface Society (TFOS) "is a condition characterized by episodic or persistent adverse ocular sensations related to lens wear, either with or without visual disturbance, resulting from reduced compatibility between the CL and the eye's environment, which can lead to decreased wearing time and discontinuation of CL wear." TFOS further states that CLD is a multifactorial condition that stems from both CL (e.g., material design, fit, care system) and environmental factors (patient factors, medication compliance, external environmental factors, ocular environment). While environmental factors related to the patient such as age and sex are inherent, rewetting drops or artificial tears can be used to treat tear film deficiencies associated with CLD. The U.S. Food & Drug Administration (FDA) defines rewetting/lubricating drops as "an in-eye solution for use with CLs" that contains "one or more active ingredients (e.g., ophthalmic demulcents) in sufficient concentration to alleviate symptoms of discomfort from CL wear by physical means." Clinicians also commonly use artificial tears off label for treating CLD and the dry eye associated with CLs because artificial tear formulations have the potential to outperform CL rewetting drops. The FDA separately classifies artificial tears as topical drops that contain specific types of demulcents or emollients. While off-label, McDonald et al. have previously shown that using a common artificial tear, Systane Ultra, before and after CL use is an effective means for treating daily disposable CL wears who have CLD. Recently, a new formulation of artificial tears, Systane Complete, was released to the market. Systane Complete is a unique formulation that has combined elements from both Systane Ultra (indicated for aqueous deficient dry eye) and Systane Balance (indicated for evaporative dry eye) to create an artificial tear with an indication for aqueous deficient, evaporative, and mixed (both aqueous deficient and evaporative) dry eye. Thus, the Research Goal of this study is to determine in a randomized clinical trial if Systane Complete is able to effectively improve the symptoms of CLD suffers.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported contact lens discomfort
* Contact Lens Dry Eye Questionnaire (CLDEQ)-8 scores ≥ 12
* Daily disposable contact lens wearer
* Best-corrected visual acuity of 20/30 or better

Exclusion Criteria:

* All other contact lens types (e.g., currently wearing two week or monthly replacement contact lenses or hard contact lenses)
* Non-compliant daily disposable contact lens wearers (must regularly replace contact lenses daily)
* Systemic health conditions known to alter tear film physiology
* History of ocular surgery within the past 12 months
* History of severe ocular trauma, active ocular infection, or inflammation
* Currently using Accutane or eye medications
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Lindenhurst Eye Physicians & Surgeons, P.C., Babylon, New York
  - Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual subject's data. Data will only be published in aggregate form.

REFERENCES:
- [Background] McDonald M, Schachet JL, Lievens CW, Kern JR. Systane(R) ultra lubricant eye drops for treatment of contact lens-related dryness. Eye Contact Lens. 2014 Mar;40(2):106-10. doi: 10.1097/ICL.0000000000000018. PMID 24552755

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Systane Complete | No Treatment
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who were 18 years an older who had a significant contact lens and dry eye questionnaire (cldeq-8) scores (12 or greater) were allowed to participate in this study. Subjects were also required to be daily disposable contact lens wearers and have a generally healthy ocular health history .
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Complete | No Treatment | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 32.7 [20 to 56] | 28.8 [18 to 69] | 30.75 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Symptoms
Description: Improvement in contact lens symptoms as measured with the Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) and CLDEQ-4 at 2 weeks compared to baseline. The CLDEQ-8 score range is 0 to 37 with 0 being the best score. Subjects were required to have a CLDEQ-8 of at least 12 in order to participate. The CLDEQ-4 is a subset of the CLDEQ-8, and it was also reported because it is a unidimensional measure of ocular discomfort in contact lens wearers. The CLDEQ-4 has a score range of 0 to 18 with 0 being the best score.
Time Frame: Baseline through 2 Weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Systane Complete | No Treatment
Number analyzed (Participants) | 22 | 24
Score on a Scale
  Baseline cldeq-8 (worse eye) | 20.41 (5.40) | 18.92 (4.92)
  2 week cldeq-8 (worse eye) | 12.86 (6.40) | 17.92 (5.30)
  Baseline cldeq-4 (worse eye) | 10.91 (3.28) | 10.38 (2.41)
  2 week cldeq-4 (worse eye) | 7.14 (3.50) | 10.13 (2.83)

2. Secondary Outcome: End of Day Eye Comfort
Description: Improvement in eye symptoms as measured with the Standardized Patient Evaluation of Eye Dryness (SPEED) at 2 weeks compared to baseline. The scale range is 0 to 28 with 0 being the best score.
Time Frame: Baseline through 2 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Systane Complete | No Treatment
Number analyzed (Participants) | 22 | 24
score on a scale
  Speed Score Baseline (worse eye) | 10.27 (3.60) | 9.67 (3.93)
  Speed Score 2 weeks (worse eye) | 7.55 (4.31) | 9.29 (4.14)

3. Secondary Outcome: Corneal Staining
Description: Improvement in conjuctivial staining at two weeks compared to baseline using the Brien Holden Vision Institute (BHVI) scale, which measures five regions of the eye on a (0-4) scale (max of 20 per metric). A score 0 is the best possible score.
Time Frame: Baseline through 2 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Systane Complete | No Treatment
Number analyzed (Participants) | 22 | 24
Units on a scale
  Corneal Staining Extent (baseline) | 1.73 (2.45) | 1.63 (2.50)
  Corneal Staining Depth (baseline) | 1.22 (1.54) | 0.92 (1.32)
  Corneal Staining Type (baseline) | 1.18 (1.56) | 0.92 (1.32)
  Corneal Staining Extent (2 weeks) | 1.41 (2.42) | 1.75 (1.98)
  Corneal Staining Depth (2 weeks) | 0.91 (1.38) | 1.04 (1.30)
  Corneal Staining Type (2 weeks) | 0.86 (1.36) | 0.92 (1.06)

4. Secondary Outcome: Schirmer's I Test Without Anesthetic
Description: Improvement in tear volume as measured in mm of wetting with a Schirmer's strip at 5 mins at 2 weeks compared to baseline. The score ranges is 0 mm to 35 mm with 35 mm being the best score.
Time Frame: Baseline through 2 Weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Systane Complete | No Treatment
Number analyzed (Participants) | 22 | 24
mm
  Schirmers Strip Baseline | 15.68 (9.70) | 20.88 (10.65)
  Schirmers Strip (2 weeks) | 15.41 (9.29) | 18.30 (10.69)

5. Secondary Outcome: Tear Break-Up Time (TBUT)
Description: Improvement in tear break up time as measured with a slit-lamp biomicroscope and sodium fluorescein in seconds at 2 weeks compared to baseline. Scores range for 0 to 60 seconds with 60 seconds being the best score.
Time Frame: Baseline through 2 Weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Systane Complete | No Treatment
Number analyzed (Participants) | 22 | 24
Seconds
  Tear Break Up Time (seconds) (baseline) | 7.70 (5.20) | 8.50 (5.10)
  Tear Break Up Time (seconds) (2 weeks) | 8.57 (4.73) | 8.80 (5.08)

ADVERSE EVENTS:
Time Frame: Data was collected 14-17 days after the baseline visit.
Description: There were no adverse events in this study
Arm/Group | Systane Complete | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

LIMITATIONS AND CAVEATS:
The results presented in this record have no known limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03682809/Prot_SAP_ICF_000.pdf